CLINICAL TRIAL: NCT01973894
Title: Whole Body Physiologically Based Pharmacokinetic (PBPK) Model to Estimate Cerebral and Systemic Midazolam Concentrations in ICU Patients Under Sedation.
Brief Title: Midazolam Whole Body Physiologically Based Pharmacokinetic Model
Acronym: MidPBPK
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Severgnini, Prof., Università degli Studi dell'Insubria
Other Study IDs: 724
Record Dates: First submitted 2012-08-19; First posted 2013-11-01 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Failure; Coma
Keywords: PBPK; Midazolam; Pharmacokinetics; Critically ill patients
MeSH Terms: conditions — Respiratory Insufficiency; Coma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Midazolam: Patients will be enrolled within 24h from the beginning of continuous Midazolam perfusion.
  Blood and urine sampling will follow this schedule:
  * 24h: blood (3ml)
  * 48h: blood (3ml) and urine
  * End of infusion: blood (3ml)
  * 6h after end of infusion: blood (3ml) and urine.
  Blood samples will be centrifuged for 10 minutes at 3300rpm, then supernatant will be placed into test tubes and stored at -20°C; urine samples will be freeze at -20°C as well.
  Then all frozen samples will be analyzed to get Midazolam concentrations.
  Interventions: Procedure: Blood and urine sampling

INTERVENTIONS:
Procedure: Blood and urine sampling — Blood and urine sampling will follow this schedule:
  * 24h: blood (3ml)
  * 48h: blood (3ml) and urine
  * End of infusion: blood (3ml)
  * 6h after end of infusion: blood (3ml) and urine. Blood samples will be centrifuged for 10 minutes at 3300rpm, then supernatant will be placed into test tubes and stored at -20°C; urine samples will be freeze at -20°C as well.
  Then all frozen samples will be analyzed to get Midazolam concentrations.

SUMMARY:
This study investigates what independent variables may influence Midazolam Pharmacokinetics in critically ill patients.

DETAILED DESCRIPTION:
This study has three specific aims:

1. to create a Midazolam PBPK model based on anthropometric and physiopathological data from enrolled patients;
2. to estimate cerebral and systemic Midazolam concentrations;
3. to assess independent variables about Midazolam pharmacokinetic in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* ICU admittance
* Caucasian
* Clinical indication of least 72h of continuous sedation with Midazolam
* MAP between 60 - 150 mmHg, even if obtained with amine support
* informed consent obtained

Exclusion Criteria:

* Any endocranial lesion, spontaneous or induced
* PaCO2 > 60 mmHg or < 30 mmHg
* PaO2 < 50 mmHg
* Pregnancy
* Anuria
* Any transplantation
* Severe hepatic failure (Child C)
* Life expectancy < 72h
* Ketoconazole and antiretrovirals in therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients in Intensive Care Unit, mechanically ventilated, sedated with midazolam, intravenous continued perfusion.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Midazolam concentration in serum and urine | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  We will calculate Midazolam AUC in serum and urine using blood and urine samples. With this data we will evaluate the elimination constants and create a Physiologically Based Pharmacokinetic Model for Midazolam simulating the drug concentration profile in brain and fat tissue.
  The blood and urine samples timing is:
  * 1 blood sample will be gathered after 24h at the beginning of continuous intravenous infusion of Midazolam
  * 1 blood sample and 1 urine sample will be gathered after 48h at the beginning of continuous intravenous infusion of Midazolam
  * 1 blood sample will be gathered at the end of continuous intravenous infusion of Midazolam (the duration of infusion is different for each patient according with clinical case)
  * 1 blood sample and 1 urine sample will be gathered after 6h at the end of continuous intravenous infusion of Midazolam (the duration of infusion is different for each patient according with clinical case)

SECONDARY OUTCOMES:
Fat mass analysis and its importance in drug distribution. | At enrollment
  At enrollment we will collect data about fat mass in our population. Our goal is to determine how much this variable can modify the distribution of Midazolam in the body. Statistical analysis will performed to found if different body mass values are correlated with different blood concentration of Midazolam at steady level.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Severgnini, Prof., Principal Investigator — Università degli Studi dell'Insubria, Varese, Italy
Locations (1):
- Azienda Ospedaliera Ospedale di Circolo e Fondazione Macchi, Varese, Italy